CLINICAL TRIAL: NCT06948630
Title: Change in Hemogram-Derived Ratios With Sepsis Filters:A Retrospective Cohort Study in the Intensive Care Unit
Brief Title: Hemogram Parameter Changes With Sepsis Filter
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: Istinye University
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Platelet Abnormality; Renal Failure; Immune System Disorder
MeSH Terms: conditions — Blood Platelet Disorders; Renal Insufficiency; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemodiafiltration is initiated in hemodynamically unstable patients in intensive care units. In some patients, additional devices called cytokine filters or sepsis filters are added to remove inflammatory cytokines. Data obtained from hemograms, such as platelet lymphocytosis ratio, are used in the diagnosis or prognosis of many diseases. This study focuses on the change in hemogram rates in patients who received hemofiltration and sepsis filters.

ELIGIBILITY:
Inclusion Criteria:

* Data of patients who were monitored in the Intensive Care between January 2020 and December 2022 and who were applied sepsis filters

Exclusion Criteria:

* -Patients who underwent hemodiafiltration with sepsis filter but could not be followed for 72 hours (death, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodiafiltration is started on patients in intensive care units. This study focuses on the change in hemogram rates in patients who underwent hemofiltration and had sepsis filters placed.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Platelet lymphocyte ratio change | up to 72 hours
  Change in platelet lymphocyte ratio measured from hemogram at the beginning (day 0) and the ratio calculated from the sample taken on day 3 in patients undergoing hemodiafiltration with sepsis filter

SECONDARY OUTCOMES:
change in the other ratios derived from complete blood cell count | up to 72 hours
  Changes in hemogram derivation ratios measured from the hemogram at the beginning (day 0) and the ratio calculated from the sample taken on day 3 in patients who underwent hemodiafiltration with sepsis filter

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Bayram, Study Chair — Istınye university faculity of Medicine
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nassiri AA, Schneider A, Hakemi MS, Sabaghian T, Ahmadi Koomleh A, Miri MM, Entezarmahdi K, Yousefzad T, Kashani K. Scientia et Cura: Illuminating the Dark Side of CRRT for Optimal Patient Benefits. Iran J Kidney Dis. 2025 Feb 25;19(1):50-58. PMID 40056440
- [Result] Wu D, Qin H. Diagnostic and prognostic values of immunocyte ratios in patients with sepsis in the intensive care unit. J Infect Dev Ctries. 2023 Oct 31;17(10):1362-1372. doi: 10.3855/jidc.17907. PMID 37956370